CLINICAL TRIAL: NCT06716840
Title: Remimazolam Besylate Versus Propofolfor Sedation of Postcardioperative Patients in Intensive Care Unit: a Prospective,Single-center,Randomized Non-inferior Trial
Brief Title: Remimazolam Besylate in Sedation of Postcardioperative Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-143
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-11

CONDITIONS: Remimazolam; Propofol; Sedation; Mechanical Ventilation; Intensive Care; Cardiac Surgery
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental)
  Interventions: Drug: Remimazolam
- propofol group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — participants in the remimazolam group received remimazolam besylate intravenously at an initial infusion rate of 0.2mg/kg/h and adjusted (maximum of 2 mg/kg/h) to maintain a Richmond Agitation-Sedation Scale(RASS) score between - 2 and 0.If the maximum dose of remimazolam was insufficient to sedate, add rescue dexmedetomidine.
  Arms: Remimazolam group
Drug: Propofol — participants in the propofol group received propofol intravenously at an initial infusion rate of 1 mg/kg/h and adjusted (maximum of 4 mg/kg/h) to maintain a Richmond Agitation-Sedation Scale (RASS) score between - 2 and 0.If the maximum dose of propofol was insufficient to sedate, add rescue dexmedetomidine.
  Arms: propofol group

SUMMARY:
Intensive care medicine is vital in managing patients after cardiac surgery with endotracheal intubation，in order to provide extensive monitoring to assure clinical stabilization. During this time of recovery, sedation is frequently employed. However, prolonged sedation risks negative sequelae.At present,propofol, benzodiazepines, and dexmedetomidine are typical drugs used for sedation of patients in intensive care unit.Each has its own advantages and disadvantages.The investigators try to find near-ideal agents for sedation,characterized by good sedative effect,minimal adverse effects and rapid awakening facilitating earlier extubation.Remimazolam appeared to be an effective and safe sedative for short term sedation. Study participants were predicated on age (> 18 years), admission following cardiac surgery, still mechanical ventilation within 48 hours,and prior informed consent.Participants were randomized to receive remimazolam besylate or propofol in a 1:1 ratio for sedation with a target sedation depth before extubation.Finally，the investigators will compare the sedation effect and safety between the 2 groups ，to prove if remimazolam is appropriate for sedation in patients after cardiac surgery in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years ;
2. admitted to the intensive care unit after cardiac surgery with techanical ventilation；
3. expected to extubation within 48hours ；
4. participant has given informed consent

Exclusion Criteria:

1. pregnant or lactating women
2. known or suspected hypersensitivity to the study drug
3. history of impaired consciousness or psychiatric illness
4. severe bradycardia with a heart rate of < 50 beats per minute
5. systolic blood pressure < 90 mmHg with fluid resuscitation and vasopressor maintenance
6. atrioventricular block（II or III degree）, Left ventricular ejection fraction(LVEF) <30%
7. participated in other clinical studies within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
percentage of time in the target sedation range | up to 2 days
  The primary outcome was the percentage of time in the target sedation range without rescue sedation.

SECONDARY OUTCOMES:
extubation time | up to 2 days
  from stopping sedative medication to removing the endotracheal tube
extubation success rate | up to 4 days
  no re-intubation within 48 hours after extubation
changes in blood pressure | up to 2 days
  dynamic changes of blood pressure were recorded during sedation
changes in heart rate | up to 2 days
  dynamic changes of heart rate were recorded during sedation
ventilator-free days | From enrollment to 7 days
  ventilator-free days at day 7
the score of confusion assessment method for the intensive care unit ( CAM-ICU) | From enrollment to the end of treatment at 28 days
  diagnose the delirium by the CAM-ICU score，and calculate the incidence of delirium
stay length | From enrollment to the end of treatment at 28 days
  length of intensive care unit stay and hospital stay
28-day mortality | From enrollment to the end of treatment at 28 days
  28-day mortality after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- First afflilated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: After the study results are published
Access Criteria: You can explain the reason and contact the study initiator via email to request the data. The email address is:yuwenqiao1980@zju.edu.cn